CLINICAL TRIAL: NCT04193592
Title: Pirfenidone in the Treatment of Hermansky Pudlak Syndrome (HPS) - Related Interstitial Lung Disease (ILD)
Brief Title: Efficacy and Safety of Pirfenidone Treatment in HPS-ILD
Acronym: PEARL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jesse Roman (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jesse Roman, Professor of Medicine, Thomas Jefferson University
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14172/2019
Record Dates: First submitted 2019-11-06; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Hermansky Pudlak Syndrome; Interstitial Lung Disease
Keywords: safety; efficacy; patient reported outcomes
MeSH Terms: conditions — Hermanski-Pudlak Syndrome; Lung Diseases, Interstitial | interventions — pirfenidone

STUDY DESIGN:
Intervention Model Description: open label drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral Pirfenidone 2403 mg per day (Experimental): Enrolled subjects will receive oral pirfenidone 801 mg taken three times a day. Pirfenidone will be supplied in 267 mg capsules.
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone will be titrated over 14 days, as tolerated, to the full dose of 2403 mg per day, as follows: Days 1 - 7: one capsule TID; Days 8 - 14: two capsules TID; Days 15 to week 52: three capsules TID. Dose may be reduced to manage an adverse event.
  Other Names: Esbriet

SUMMARY:
This research study will explore the safety and efficacy of the drug, pirfenidone, in patients with a diagnosis of Hermansky-Pudlak Syndrome (HPS) who have an associated interstitial lung disease (ILD) over a planned period of 56 weeks.

DETAILED DESCRIPTION:
An open-label clinical study designed to evaluate the efficacy and safety of administering pirfeniodne for 52 weeks to subjects with HPS-ILD. Patients meeting the eligibility criteria without contraindications for the study will be provided pirfenidone 2403 mg/day. Efficacy will be evaluated through interval testing of pulmonary function tests, patient reported outcomes, adverse events and survival. Safety will be assessed by determining adverse events, hospitalizations, and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Probable or definite diagnosis of HPS based on confirmed genetic mutation or clinical picture characterized by oculo-cutaneous albinism, bleeding disorder, and possible colitis and ILD.
* Diagnosis of ILD supported by clinically indicated HRCT prior to Screening, and presence of fibrotic abnormality affecting more than 5% of the lung parenchyma, with or without traction bronchiectasis or honeycombing, on Screening
* No features supporting an alternative diagnosis (e.g., infection)
* Change in pre-bronchodilator FVC (measured in liters) between Screening (Visit 1) and

Baseline (Visit 2) must be a < 10% relative difference, calculated as:

100%*[absolute value (Screening FVC - Baseline FVC)/Screening FVC

* Stable dose (at least three months at the time of Screening) of corticosteroids.
* No cytotoxic, immunosuppresive agents, cytokine-modulating, or receptor antagonists agents are allowed (including but not limited to azathioprine, cyclophosphamide, cyclosporine, etanercept, iloprost, infliximab, methotrexate, mycophenolate mofetil, nintedanib, tacrolimus, tetrathiomolybdate, TNF-α inhibitors, rituximab, abatacept, tofacitintib, tociluzimab).
* Able to understand and sign a written informed consent form

Exclusion Criteria:

* Not a suitable candidate for enrollment or unlikely to comply with the requirements of this study, in the opinion of the investigator
* Cigarette smoking within 3 months of Screening or unwilling to avoid tobacco products throughout the study
* History of clinically significant environmental exposure known to cause pulmonary fibrosis (PF), including but not limited to drugs (such as amiodarone), asbestos, beryllium, radiation, and domestic birds
* Concurrent presence of other interstitial lung disease, including but not limited to radiation, drug toxicity, sarcoidosis, hypersensitivity pneumonitis, bronchiolitis obliterans organizing pneumonia, human immunodeficiency virus (HIV), viral hepatitis, and cancer
* Concurrent presence of other pleuropulmonary manifestations inconsistent with HPS- ILD
* Presence of pleural effusion occupying more than 10% of the hemithorax on Screening HRCT
* Clinical diagnosis of a connective tissue disease or overlap syndrome (including but not limited to rheumatoid arthritis, scleroderma, polymyositis/dermatomyositis, systemic lupus erythematosus)
* Coexistent clinically significant COPD/emphysema or asthma in the opinion of the site principle investigator
* Clinical evidence of active infection, including but not limited to bronchitis, pneumonia, sinusitis, urinary tract infection, or cellulitis
* Any history of malignancy diagnosed within 5 years of screening, other than basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or low grade cervical carcinoma in situ.
* History of severe hepatic impairment or end-stage liver disease
* History of end-stage renal disease requiring dialysis
* History of unstable or deteriorating cardiac or disease, myocardial infarction within the previous year, heart failure within the last 3 years, or cardiac arrhythmia requiring drug therapy
* Any condition that, in the opinion of the investigator, might be significantly exacerbated by the known side effects associated with the administration of pirfenidone
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use two adequate methods of contraception, including at least one method with a failure rate of <1% per year, during the 52 weeks of treatment.

  1. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
  2. Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, established and proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  3. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* For men who are not surgically sterile: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

  1. With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 118 days after the last dose of pirfenidone.
  2. Men must refrain from donating sperm during this same period.
* Investigational therapy, defined as any drug that has not been approved for marketing for any indication in the country of the participating site including pirfenidone, at the time of Screening
* History of alcohol or substance abuse in the past 2 years, at the time of Screening
* Family or personal history of long QT syndrome
* Any of the following liver function test criteria above specified limits:

  1. Total bilirubin above the upper limit of normal (ULN), excluding patients with Gilbert's syndrome; aspartate or alanine aminotransferase (AST/SGOT or ALT/SGPT) >3 × ULN; alkaline phosphatase >2.5 × ULN
  2. Creatinine clearance (CrCl <30) mL/min, calculated using the Cockcroft-Gault formula
  3. Electrocardiogram (ECG) with a QTcB interval >500 msec at Screening
* Prior use of pirfenidone or known hypersensitivity to any of the components of study treatment
* Use of any of the following therapies within 28 days before Screening:

  1. Investigational therapy, defined as any drug that has not been approved for marketing for any indication in the country of the participating site
  2. Fluvoxamine
  3. Sildenafil (daily use). Note: intermittent use for erectile dysfunction is allowed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Forced Vital Capacity (FVC) | baseline, 6 months, 12 months
  The incidence of decline in percent predicted FVC of 10 % or greater from baseline measured at 6 and 12 months

SECONDARY OUTCOMES:
Change in Forced Vital Capacity (FVC) | week 52
  1. The Incidence of decline from baseline in percent predicted FVC of 10% or greater during the 52 week treatment period.
Change in Diffusion Capacity (DLCO) | week 52
  2. The Incidence of decline from baseline in percent predicted DLCO of 15% or greater during the 52 week treatment period.
Incidence of Treatment Emergent Adverse Events | week 52
  3. The number of participants with and number of treatment emergent adverse events reported by the participant will be collected.
Incidence of Treatment Emergent Serious Adverse Events | week 52
  4. The number of participants with and number of treatment-emergent serious adverse events reported by the participants will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Roman, MD, Principal Investigator — Thomas Jefferson University
Locations (2):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States
- Mayaguez Medical Center, Mayagüez, Puerto Rico

IPD SHARING:
Plan to Share IPD: No